CLINICAL TRIAL: NCT04953767
Title: The Circadian Rhythm of ICU Patients With Acute Myocardial Infraction and the Effect of Dynamic Light Therapy : A Preliminary Study
Brief Title: The Circadian Rhythm of ICU Patients With Acute Myocardial Infraction and the Effect of Light Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201902108A3
Record Dates: First submitted 2021-06-21; First posted 2021-07-08 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Circadian Dysrhythmia; Delirium
Keywords: Circadian rhythm; ICU; Acute myocardial infarction; Delirium; Light therapy
MeSH Terms: conditions — Delirium | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blue light therapy (Experimental): The participants receive blue light therapy for 1 hours, between 8am to 12pm in the morning.
  Interventions: Device: Blue light therapy
- White light (Sham Comparator): The participants receive white light for 1 hour, between 8am to 12pm in the morning.
  Interventions: Other: White light

INTERVENTIONS:
Device: Blue light therapy — Blue light therapy has been proved its efficacy and safety is treatment circadian rhythm disorder as well as other diseases.
  Arms: Blue light therapy
Other: White light — White light is used as sham control.
  Arms: White light

SUMMARY:
By using subjective and objective measurements, the investigators monitor the change of circadian rhythm in Intensive Care Unit (ICU) patients with acute myocardial infarction and the effect of light therapy.

DETAILED DESCRIPTION:
The investigators include 70 patients who are admitted to coronary care unit due to coronary artery disease, with severity between Killip I-III and age between 35-85. Participants are randomly assigned to 2 groups, the experimental group (blue light) and the placebo group (white light). Both groups receive light therapy or white light daily between 8am to 12pm. The investigators use actigraphy and heart rate variation analysis, and check melatonin level as objective measurements. The investigators use delirium scales to evaluate delirium and its severity. The light therapy is stopped once a participant is diagnosed of delirium or transferred, and the investigators keep following participants until discharge to evaluate the prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis for admission is acute myocardial infarction with severity between Killip I-III.
* Age is between 35-85.
* Participants who are willing to participate in the study and sign the informed consent.

Exclusion Criteria:

* Using sedative hypnotic drugs.
* Blindness or severe cataract.
* Neurological diseases such as epilepsy, brain injury, or stroke.
* Severe mental disorder such as major depressive disorder, bipolar disorder, schizophrenia, intellectual disability or substance use disorders.
* Unable to communicate.
* Participants who are unwilling to participate in the study or refuse to sign the informed consent.
* Participants who are not suitable to include in this study, evaluate by PI or Co-PI.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes of the circadian rhythm during admission by actigraphy | an average of 2 weeks of continuous monitoring since baseline till discharge, up to 4 weeks
  Actigraphy data
Changes of the circadian rhythm during admission by heart-rate-variation-analysis | baseline for 48hours, and 24hours before discharge
  heart-rate-variation-analysis data
Changes of Melatonin level | collect saliva in the morning and at the night of Day 1 and the day of discharge
  Melatonin level
Changes of Vitamin D level | blood sampling at Day 1 and the day of discharge
  Vitamin D level

SECONDARY OUTCOMES:
Confusion Assessment Method for the Intensive Care Unit | evaluate daily since baseline to discharge, for an average of 2 weeks, up to 4 weeks
  Evaluation of delirium and its severity, score range 0-7, and score 0-2 no delirium, 3-5 mild to moderate, 6-7 severe
Intensive Care Delirium Screen Checklist | evaluate daily since baseline to discharge, for an average of 2 weeks, up to 4 weeks
  Evaluation of delirium and its severity, score range 0-8, and score 4-8 suspected delirium

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chih Chin, Principal Investigator — Chang Gung Medical Foundation
Locations (1):
- Wei-Chih Chin, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salluh JI, Wang H, Schneider EB, Nagaraja N, Yenokyan G, Damluji A, Serafim RB, Stevens RD. Outcome of delirium in critically ill patients: systematic review and meta-analysis. BMJ. 2015 Jun 3;350:h2538. doi: 10.1136/bmj.h2538. PMID 26041151
- [Background] van Maanen A, Meijer AM, van der Heijden KB, Oort FJ. The effects of light therapy on sleep problems: A systematic review and meta-analysis. Sleep Med Rev. 2016 Oct;29:52-62. doi: 10.1016/j.smrv.2015.08.009. Epub 2015 Sep 9. PMID 26606319
- [Background] Ono H, Taguchi T, Kido Y, Fujino Y, Doki Y. The usefulness of bright light therapy for patients after oesophagectomy. Intensive Crit Care Nurs. 2011 Jun;27(3):158-66. doi: 10.1016/j.iccn.2011.03.003. Epub 2011 Apr 21. PMID 21511473
- [Background] Taguchi T, Yano M, Kido Y. Influence of bright light therapy on postoperative patients: a pilot study. Intensive Crit Care Nurs. 2007 Oct;23(5):289-97. doi: 10.1016/j.iccn.2007.04.004. Epub 2007 Aug 9. PMID 17692522
- [Background] Oh J, Cho D, Park J, Na SH, Kim J, Heo J, Shin CS, Kim JJ, Park JY, Lee B. Prediction and early detection of delirium in the intensive care unit by using heart rate variability and machine learning. Physiol Meas. 2018 Mar 27;39(3):035004. doi: 10.1088/1361-6579/aaab07. PMID 29376502
- [Background] Osse RJ, Tulen JH, Hengeveld MW, Bogers AJ. Screening methods for delirium: early diagnosis by means of objective quantification of motor activity patterns using wrist-actigraphy. Interact Cardiovasc Thorac Surg. 2009 Mar;8(3):344-8; discussion 348. doi: 10.1510/icvts.2008.192278. Epub 2008 Dec 22. PMID 19103609
- [Background] Papaioannou VE, Maglaveras N, Houvarda I, Antoniadou E, Vretzakis G. Investigation of altered heart rate variability, nonlinear properties of heart rate signals, and organ dysfunction longitudinally over time in intensive care unit patients. J Crit Care. 2006 Mar;21(1):95-103; discussion 103-4. doi: 10.1016/j.jcrc.2005.12.007. PMID 16616632